CLINICAL TRIAL: NCT07029464
Title: Comparison of Short- and Long-term Outcomes Between Robotic and Laparoscopic Hemicolectomy of Right Colon Cancer : A Multicenter Propensity Score Matching Analysis
Status: Not yet recruiting | Type: Observational
Sponsor: The First Affiliated Hospital of Nanchang University (Other)
Collaborators: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); Fudan University (Other); The Second Affiliated Hospital of Harbin Medical University (Other); Three Gorges Hospital of Chongqing University (Other); The Affiliated Hospital of Qingdao University (Other); The First Affiliated Hospital of Zhengzhou University (Other); Tianjin Third Central Hospital (Other); Shandong University Second Hospital (Unknown); Nanfang Hospital, Southern Medical University (Other); Huadong Hospital (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Second Xiangya Hospital of Central South University (Other); Jiangxi Provincial People's Hopital (Other); Pingxiang People 's Hospital (Unknown); Ganzhou City People's Hospital (Other)
Responsible Party: Principal Investigator, Taiyuan Li, chief physician, The First Affiliated Hospital of Nanchang University
Other Study IDs: IITS2025462
Record Dates: First submitted 2025-05-26; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Robotic Surgical Procedures; Right Colon Tumors; Cancer; Laparoscopic Abdominal Surgery
Keywords: right colon cancer; robotic surgery
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- R Group: robotic surgery
- L Group: Laparoscopic surgery

SUMMARY:
This is a retrospective, multicenter cohort study to compare short- and long-term outcomes between robotic and laparoscopic hemicolectomy of right colon cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1.Underwent radical right hemicolectomy by Da Vinci robotic or laparoscopic surgery 2.Postoperative pathology confirmed right colon adenocarcinoma (pT2-T4aNxM0; including cecal adenocarcinoma, ascending colon adenocarcinoma, hepatic flexure colon adenocarcinoma, and proximal transverse colon adenocarcinoma) 3.Complete clinical data and pathological results available

Exclusion Criteria:

* 1.Received neoadjuvant therapy prior to surgery 2.History of other malignancies in the past 5 years (except cured cervical carcinoma in situ, basal cell carcinoma, or squamous cell carcinoma of the skin) 3.Distant metastases (e.g., liver, lung) or extensive abdominal/pelvic metastases confirmed by contrast-enhanced CT, PET-CT, or intraoperative exploration 4.Comorbid neurological/psychiatric disorders impairing ability to express informed consent 5.Poor systemic condition with contraindications to general anesthesia 6.Severe obesity (BMI >35 kg/m²) 7.Severe widespread abdominal adhesions precluding safe pneumoperitoneum establishment 8.Emergency surgery due to tumor perforation or obstruction 9.Refusal to provide informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The procedures were performed by 16 surgeons from 16 participating centers. Both primary surgeons and assistants completed standardized training in robotic and laparoscopic surgical techniques and obtained certification. Each center performs over 100 robotic- or laparoscopic-assisted radical right hemicolectomies annually. Primary surgeons had performed at least 50 cases of both robotic and laparoscopic-assisted radical right hemicolectomy.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
3-year overall survival (OS) rate and 3-year disease-free survival (DFS) rate | （OS）From post-operation until death or the 3-year study endpoint （DFS）From post-operation to tumor recurrence or the 3-year study endpoint

SECONDARY OUTCOMES:
Operative time | Periprocedural
Intraoperative blood loss | Periprocedural
Time to first flatus/bowel movement | Periprocedural
Time to liquid diet initiation | Periprocedural
Time to ambulation | Periprocedural
Postoperative hospital stay duration | Up to 30 days
Postoperative complications | From end of surgery to 30 days postoperatively
  Surgery-related adverse events within 30 days, graded via the Clavien-Dindo classification system
Postoperative white blood cell (WBC) count | On postoperative days 1, 3, and 5
  Measured on postoperative days 1, 3, and 5
Postoperative C-reactive protein (CRP) level | On postoperative days 1, 3, and 5
  Measured on postoperative days 1, 3, and 5
Pain score | On postoperative days 1, 3, and 5
  Assessed using the Visual Analog Scale (VAS) on postoperative days 1, 3, and 5

IPD SHARING:
Plan to Share IPD: No